CLINICAL TRIAL: NCT05012826
Title: Osteopathy and Physiotherapy Compared to Physiotherapy Alone on Fatigue and Functional Status in Long COVID: Study Protocol for a Pragmatic Randomized Controlled SuperiorityTrial
Brief Title: Osteopathy and Physiotherapy Compared to Physiotherapy Alone on Fatigue and Functional Status in Long COVID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centro Universitário Augusto Motta (Other)
Collaborators: Instituto Brasileiro de Osteopatia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38342520.7.0000.5235
Record Dates: First submitted 2021-08-16; First posted 2021-08-19 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Covid19; SARS-CoV-2 Infection
Keywords: COVID-19; SARS-CoV-2; Physical Therapy Modalities; Osteopathic Manipulation; Rehabilitation
MeSH Terms: conditions — COVID-19 | interventions — Manipulation, Osteopathic; Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Two-arm, controlled, assessor-blinded, pragmatic randomized controlled superiority trial
Who Masked: Outcomes Assessor
Masking Description: To ensure the expectation of treatment is equally balanced between the groups the participants will not be aware of the study hypothesis regarding the between-group comparisons. It is not possible to blind the clinicians regarding the groups and the participants regarding their treatment. The outcome assessor and statistician will be blind to the allocations of groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Osteopathic Manipulative Treatment (OMT)+ Physiotherapy (PT) Group (Experimental): Participants in this group will receive OMT in addition to the same interventions of PT group for the same 2- month period. The frequency of treatment will be decided based on the clinical judgment of the osteopath who is accompanying each case, not exceeding 7 consultations in total. At each visit, the participants will receive a full-body osteopathic examination which include clinical exams, observation, screening tests, palpation, and motion testing. The OMT entail direct (high-velocity low-amplitude; muscle energy; and myofascial release), indirect (functional techniques and balanced ligamentous tension), visceral, and cranial techniques(Giusti, 2017). Selection of specific OMT will follow the 'TART' criteria-Tissue texture changes, Asymmetry, Restriction of motion, Tenderness (Basile et al., 2017; Cerritelli et al., 2011; Giusti R., 2017; Pizzolorusso et al., 2011; Seffinger M.A, 2018).
  Interventions: Other: Osteopathic Manipulative Treatment in addition to Physiotherapy; Other: Physiotherapy
- Physiotherapy Group (PT) (Active Comparator): Participants in this group will receive physiotherapy sessions with a maximum frequency of 2 weekly sessions, as defined by the physiotherapist, according to personalized therapeutic plans for a period of 2 months. The physiotherapy approach for patients with long COVID includes motor and respiratory rehabilitation aiming at maintaining and/or improving joint mobility, muscle strength, and functional exercise capacity (Thomas et al., 2020). At each visit, the participants respond by self-report about their general condition. Depending on the case, the physiotherapist will perform a reevaluation with specific tests. The PT group will receive physiotherapy treatment offered by five physiotherapists, with more than 5 years of experience each, duly registered with their class council. the treatment provided will be registered on each participant's clinical notes and a summary of main interventions will be reported.
  Interventions: Other: Physiotherapy

INTERVENTIONS:
Other: Osteopathic Manipulative Treatment in addition to Physiotherapy — Participants in this group will receive OMT in addition to the same interventions of PT group. The frequency of treatment will be decided based on the clinical judgment of the osteopath who is accompanying each case, not exceeding 7 consultations in total. At each visit, the participants will receive a full-body osteopathic examination which include clinical exams, observation, screening tests, palpation, and motion testing. The OMT entail direct (high-velocity low-amplitude; muscle energy; and myofascial release), indirect (functional techniques and balanced ligamentous tension), visceral, and cranial techniques(Giusti, 2017). Selection of specific OMT will follow the 'TART' criteria-Tissue texture changes, Asymmetry, Restriction of motion, Tenderness (Basile et al., 2017; Cerritelli et al., 2011; Giusti R., 2017; Pizzolorusso et al., 2011; Seffinger M.A, 2018).
  Arms: Osteopathic Manipulative Treatment (OMT)+ Physiotherapy (PT) Group
Other: Physiotherapy — Participants in this group will receive physiotherapy sessions with a maximum frequency of 2 weekly sessions, as defined by the physiotherapist, according to personalized therapeutic plans for a period of 8 weeks. The physiotherapy approach for patients with long COVID includes motor and respiratory rehabilitation aiming at maintaining and/or improving joint mobility, muscle strength, and functional exercise capacity (Thomas et al., 2020). At each visit, the participants respond by self-report about their general condition. Depending on the case, the physiotherapist will perform a reevaluation with specific tests. The PT group will receive physiotherapy treatment offered by five physiotherapists, with more than 5 years of experience each, duly registered with their class council.

SUMMARY:
Background: Fatigue is among the most common symptoms of the long-term effects of coronavirus (long COVID). This study aims to compare the effectiveness of osteopathic manipulative treatment (OMT) combined with physiotherapy treatment (PT) compared to PT alone on fatigue and functional limitations after two months post randomization in adults with long COVID.

Methods: This is a study protocol for a two-arm, assessor-blinded, pragmatic randomized controlled superiority trial. Seventy-six participants will be randomly allocated to OMT+PT or PT. The PT includes usual care interventions including motor and respiratory exercises targeting cardiorespiratory and skeletal muscle functions. The OMT entails direct, indirect, visceral, and cranial techniques. Patients will be evaluated before and after a 2-month intervention program, and at 3-month follow-up session. Primary objectives comprise fatigue and functional limitations at 2-month post randomization as assessed by the fatigue severity scale and the Post-COVID Functional State scale. Secondary objectives comprise fatigue and functional limitations at 3 months, and the perceived change post-treatment as assessed by the Perceived Change Scale (PCS-patient).

DETAILED DESCRIPTION:
The coronavirus disease caused by the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)-COVID-19-is causing a substantial increase in hospitalizations leading to overloads in global health systems. Long-term effects of coronavirus-long COVID-comprise of the effects of COVID-19 that lasts for weeks or even months beyond the acute infection. Long COVID includes a wide spectrum of respiratory, neurologic, cardiovascular, gastrointestinal, and musculoskeletal symptoms, and an increased risk of death. There are more than 50 known possible sequelae in long COVID, such as chronic fatigue, and the clinical manifestations may persist for weeks after the acute infection [6], leading to a decrease in quality of life. This condition reinforces the demand for healthcare and the need for a comprehensive approach for patients with long COVID.

Physiotherapy interventions may be required for patients with long COVID aiming to manage symptoms, prevent and restore the patients' functional status and enabling them to perform activities of daily living. The physiotherapy approach for patients with long COVID includes motor and respiratory rehabilitation aiming at maintaining and/or improving joint mobility, muscle strength, and functional capacity. A systematic review highlighted that to improve the rehabilitation in patients, especially in older adults with a severe respiratory illness on admission and after post ICU, some exercise regimens and habits can bring hope, confidence, and functional independence. The authors suggest this may be generalized to those treated for COVID-19, but maybe with personalized care. However, there is a lack of consensus on outcomes measures.

Osteopathy is a healthcare system that aims to promote the balance of physiological function, support homeostasis and encourage wellbeing. In 1918, during the Spanish flu in the United States, osteopathy presented itself as one of the health resources made available to help fight the epidemic. In 2007, OMT once again presented itself as a possibility to help restore health to individuals affected by the H5N1 avian flu. It is worth noticing though these studies are of the lowest evidence, often collections of research that is not directly relevant to the condition and with no indication of clinical relevance; also, most of them comprise hypothetical opinions on this matter. Studies on the OMT combined with standard medical care show that OMT can collaborate in the recovery of health in various clinical conditions, including shortening the length of stay and in-hospital mortality rates in the elderly with more severe pneumonia. Altogether, the interest in the field but absence of reliable data justified an effort to assess the effects of OMT on fatigue in people with long COVID. If found effective, OMT may be recommended as an adjunct to other interventions for this population.

Fatigue is one of the most common and persistent sequelae in long COVID. Fatigue is often a disabling symptom related to several clinical conditions related to systemic inflammatory processes. Pain and fatigue, for example, may overlap, suggesting that biological mechanisms, which include peripheral and central components, and identifiable neuronal networks, are present in both conditions. In a systematic review of the effects of OMT on chronic inflammatory diseases, the data proved inconsistent but safe, suggesting more robust trials are warranted. Hence, the primary aim of this trial is to test whether OMT combined with PT (OMT+PT) is superior to PT alone on fatigue and functional limitations two months post randomization in adults with long COVID. Secondarily, this trial will investigate the effectiveness of OMT+PT and PT alone on fatigue, functional status, and perceived change post-treatment 3 months post-randomization in this population.

ELIGIBILITY:
Inclusion Criteria: comprise age equal to or above 18 years; essential and clinical criteria for long COVID at baseline assessment (confirmed preceding infection with SARS-CoV-2, individuals referred for rehabilitation reporting fatigue as major symptom [35]; and ability to understand Portuguese well enough to be able to fill in the questionnaires

Exclusion Criteria: comprise conditions in which fatigue is also a major complain such as suspected or diagnosed chronic and/or neurological diseases (e.g., Parkinson's disease, amyotrophic lateral sclerosis, Alzheimer's disease); pre-existing, chronic diseases affecting the musculoskeletal system (e.g., fibromyalgia).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2021-09-20 (Actual); Primary Completion 2023-06-06 (Estimated); Study Completion 2023-07-06 (Estimated)

PRIMARY OUTCOMES:
Fatigue | 90 days
  Fatigue Severity Scale: the scale consists of 9 items on how fatigue interferes with certain activities. Severity is classified according to a self-report scale. The scale consists of a 7-point score where 1 = strongly disagree and 7 = strongly agree. The minimum score is 9 and the maximum is 63. The higher the score is the greater the severity of fatigue (Krupp et al., 1989; Toledo et al., 2011). The Portuguese-Brazil version of FSS has high reliability (Cronbach's alpha = 0.93) and good construct validity with pain and fatigue instruments (Pearson correlation of 0.60 and 0.56, respectively)
Functional status | 90 days
  The Post-COVID Functional State Scale : The scale has a score from 0 to 4 with 0 being no functional limitation and 4 severe functional limitation. In the present study, we will use the patient's flowchart and questionnaire with translation into Portuguese language (https://osf.io/qgpdv/) regarding his condition on the day of application (Klok et al., 2020).The Portuguese-Brazil version of PCFS has weak-to-strong construct validity (Pearson correlation in range 0.233 to 0.661) with health-related quality of life

SECONDARY OUTCOMES:
Global impression of recovery | 90 days
  The Perceived Change Scale (Patient Version): . It has 19 items, 18 of which assess the perceived changes related to: occupation and physical health, psychological dimension and sleep, relationships, and emotional stability, in addition to a last item that globally assesses the perceived change. Each item has 3-point Likert responses, where point 1 equates to worse than before, 2 to no change and 3 to better than before (Bandeira et al., 2011; Perreault et al., 2010).than before [43]. The Portuguese-Brazil version of EMP-patient has good internal consistency (Cronbach alpha = 0.85), test-retest temporal stability (Pearson correlation = 0.93) and convergent construct validity with a service satisfaction instrument (Pearson correlation = 0.37)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Christina Ce Curi, MsC, Principal Investigator — Centro Universitário Augusto Motta
Locations (1):
- Hospital Municipal de Reabilitação de Engenho de dentro, Rio de Janeiro, Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Adams J, Sibbritt D, Steel A, Peng W. A workforce survey of Australian osteopathy: analysis of a nationally-representative sample of osteopaths from the Osteopathy Research and Innovation Network (ORION) project. BMC Health Serv Res. 2018 May 10;18(1):352. doi: 10.1186/s12913-018-3158-y. PMID 29747647
- [Background] Altman DG, Schulz KF, Moher D, Egger M, Davidoff F, Elbourne D, Gotzsche PC, Lang T; CONSORT GROUP (Consolidated Standards of Reporting Trials). The revised CONSORT statement for reporting randomized trials: explanation and elaboration. Ann Intern Med. 2001 Apr 17;134(8):663-94. doi: 10.7326/0003-4819-134-8-200104170-00012. PMID 11304107
- [Background] Alvarez G, Roura S, Cerritelli F, Esteves JE, Verbeeck J, van Dun PLS. The Spanish Osteopathic Practitioners Estimates and RAtes (OPERA) study: A cross-sectional survey. PLoS One. 2020 Jun 15;15(6):e0234713. doi: 10.1371/journal.pone.0234713. eCollection 2020. PMID 32542047
- [Background] Costa CS, Bandeira M, Cavalcanti RL, Scalon JD. [Perceptions by patients and families towards treatment outcomes in mental health services]. Cad Saude Publica. 2011 May;27(5):995-1007. doi: 10.1590/s0102-311x2011000500017. Portuguese. PMID 21655850
- [Background] Basile, F., Scionti, R., & Petracca, M. (2017). Diagnostic reliability of osteopathic tests: A systematic review. International Journal of Osteopathic Medicine, 25, 21-29. https://doi.org/10.1016/j.ijosm.2017.03.004
- [Background] Bordoni B, Zanier E. Understanding Fibroblasts in Order to Comprehend the Osteopathic Treatment of the Fascia. Evid Based Complement Alternat Med. 2015;2015:860934. doi: 10.1155/2015/860934. Epub 2015 Aug 19. PMID 26357524
- [Background] Cerritelli F, Carinci F, Pizzolorusso G, Turi P, Renzetti C, Pizzolorusso F, Orlando F, Cozzolino V, Barlafante G. Osteopathic manipulation as a complementary treatment for the prevention of cardiac complications: 12-Months follow-up of intima media and blood pressure on a cohort affected by hypertension. J Bodyw Mov Ther. 2011 Jan;15(1):68-74. doi: 10.1016/j.jbmt.2010.03.005. Epub 2010 May 8. PMID 21147421
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Dal Farra F, Risio RG, Vismara L, Bergna A. Effectiveness of osteopathic interventions in chronic non-specific low back pain: A systematic review and meta-analysis. Complement Ther Med. 2021 Jan;56:102616. doi: 10.1016/j.ctim.2020.102616. Epub 2020 Nov 13. PMID 33197571
- [Background] de Zoete A, de Boer MR, Rubinstein SM, van Tulder MW, Underwood M, Hayden JA, Buffart LM, Ostelo R; International IPD-SMT group. Moderators of the Effect of Spinal Manipulative Therapy on Pain Relief and Function in Patients with Chronic Low Back Pain: An Individual Participant Data Meta-analysis. Spine (Phila Pa 1976). 2021 Apr 15;46(8):E505-E517. doi: 10.1097/BRS.0000000000003814. PMID 33186277
- [Background] van Dun P.L.S., Kouwenberg T. (red.), 2012, The Scope of Osteopathic Practice in Europe, Brussels, European Federation of Osteopaths (EFO) & Forum for Osteopathic Regulation in Europe (FORE)van Dun P.L.S., Kouwenberg T. (red.), 2012, The Scope of Osteopathic Practice in Europe, Brussels, European Federation of Osteopaths (EFO) & Forum for Osteopathic Regulation in Europe (FORE)
- [Background] Giusti, R. (2017). glossary OF OSTEOPATHIC TERMINOLOGY Third Edition.
- [Background] Goodwin VA, Allan L, Bethel A, Cowley A, Cross JL, Day J, Drummond A, Hall AJ, Howard M, Morley N, Thompson Coon J, Lamb SE. Rehabilitation to enable recovery from COVID-19: a rapid systematic review. Physiotherapy. 2021 Jun;111:4-22. doi: 10.1016/j.physio.2021.01.007. Epub 2021 Feb 24. PMID 33637294
- [Background] Health, W. H. O., Programme, E., Panel, E. A., Preparedness, I. P. C., Guidance, I. P. C., Group, D., Gdg, I. P. C., Preparedness, S., & Plan, R. (2020). Transmission of SARS-CoV-2 : implications for infection prevention precautions. July, 1-10.
- [Background] Hoffmann TC, Glasziou PP, Boutron I, Milne R, Perera R, Moher D, Altman DG, Barbour V, Macdonald H, Johnston M, Lamb SE, Dixon-Woods M, McCulloch P, Wyatt JC, Chan AW, Michie S. Better reporting of interventions: template for intervention description and replication (TIDieR) checklist and guide. BMJ. 2014 Mar 7;348:g1687. doi: 10.1136/bmj.g1687. PMID 24609605
- [Background] Hruby RJ, Hoffman KN. Avian influenza: an osteopathic component to treatment. Osteopath Med Prim Care. 2007 Jul 9;1:10. doi: 10.1186/1750-4732-1-10. PMID 17620133
- [Background] Kim L, Garg S, O'Halloran A, Whitaker M, Pham H, Anderson EJ, Armistead I, Bennett NM, Billing L, Como-Sabetti K, Hill M, Kim S, Monroe ML, Muse A, Reingold AL, Schaffner W, Sutton M, Talbot HK, Torres SM, Yousey-Hindes K, Holstein R, Cummings C, Brammer L, Hall AJ, Fry AM, Langley GE. Risk Factors for Intensive Care Unit Admission and In-hospital Mortality Among Hospitalized Adults Identified through the US Coronavirus Disease 2019 (COVID-19)-Associated Hospitalization Surveillance Network (COVID-NET). Clin Infect Dis. 2021 May 4;72(9):e206-e214. doi: 10.1093/cid/ciaa1012. PMID 32674114
- [Background] Klok FA, Boon GJAM, Barco S, Endres M, Geelhoed JJM, Knauss S, Rezek SA, Spruit MA, Vehreschild J, Siegerink B. The Post-COVID-19 Functional Status scale: a tool to measure functional status over time after COVID-19. Eur Respir J. 2020 Jul 2;56(1):2001494. doi: 10.1183/13993003.01494-2020. Print 2020 Jul. PMID 32398306
- [Background] Krupp LB, LaRocca NG, Muir-Nash J, Steinberg AD. The fatigue severity scale. Application to patients with multiple sclerosis and systemic lupus erythematosus. Arch Neurol. 1989 Oct;46(10):1121-3. doi: 10.1001/archneur.1989.00520460115022. PMID 2803071
- [Background] Lesho E, McKeown A, Laguio-Vila M. The rationale for including osteopathic manipulative treatment in the management of infections: a hermeneutic review. Expert Rev Anti Infect Ther. 2022 Jan;20(1):23-31. doi: 10.1080/14787210.2021.1935236. Epub 2021 Jun 7. PMID 34034598
- [Background] Lopez-Leon S, Wegman-Ostrosky T, Perelman C, Sepulveda R, Rebolledo PA, Cuapio A, Villapol S. More than 50 long-term effects of COVID-19: a systematic review and meta-analysis. Sci Rep. 2021 Aug 9;11(1):16144. doi: 10.1038/s41598-021-95565-8. PMID 34373540
- [Background] Marin T, Maxel X, Robin A, Stubbe L. Evidence-based assessment of potential therapeutic effects of adjunct osteopathic medicine for multidisciplinary care of acute and convalescent COVID-19 patients. Explore (NY). 2021 Mar-Apr;17(2):141-147. doi: 10.1016/j.explore.2020.09.006. Epub 2020 Sep 25. PMID 33158784
- [Background] Meltzer, K. R., & Standley, P. R. (2007). Context: Clinical studies have supported the efficacy of a variety of osteopathic manipulative techniques. However, an evidence base for the cellular mechanisms underlying these clinical findings is lacking. 107(12), 527-536.
- [Background] Muller A, Franke H, Resch KL, Fryer G. Effectiveness of osteopathic manipulative therapy for managing symptoms of irritable bowel syndrome: a systematic review. J Am Osteopath Assoc. 2014 Jun;114(6):470-9. doi: 10.7556/jaoa.2014.098. PMID 24917634
- [Background] Nalbandian A, Sehgal K, Gupta A, Madhavan MV, McGroder C, Stevens JS, Cook JR, Nordvig AS, Shalev D, Sehrawat TS, Ahluwalia N, Bikdeli B, Dietz D, Der-Nigoghossian C, Liyanage-Don N, Rosner GF, Bernstein EJ, Mohan S, Beckley AA, Seres DS, Choueiri TK, Uriel N, Ausiello JC, Accili D, Freedberg DE, Baldwin M, Schwartz A, Brodie D, Garcia CK, Elkind MSV, Connors JM, Bilezikian JP, Landry DW, Wan EY. Post-acute COVID-19 syndrome. Nat Med. 2021 Apr;27(4):601-615. doi: 10.1038/s41591-021-01283-z. Epub 2021 Mar 22. PMID 33753937
- [Background] Noll DR, Degenhardt BF, Johnson JC. Multicenter Osteopathic Pneumonia Study in the Elderly: Subgroup Analysis on Hospital Length of Stay, Ventilator-Dependent Respiratory Failure Rate, and In-hospital Mortality Rate. J Am Osteopath Assoc. 2016 Sep 1;116(9):574-87. doi: 10.7556/jaoa.2016.117. PMID 27571294
- [Background] Nordin A, Taft C, Lundgren-Nilsson A, Dencker A. Minimal important differences for fatigue patient reported outcome measures-a systematic review. BMC Med Res Methodol. 2016 May 26;16:62. doi: 10.1186/s12874-016-0167-6. PMID 27387456
- [Background] Perreault M, White ND, Fabres E, Landry M, Anestin AS, Rabouin D. Relationship between perceived improvement and treatment satisfaction among clients of a methadone maintenance program. Eval Program Plann. 2010 Nov;33(4):410-7. doi: 10.1016/j.evalprogplan.2009.12.003. Epub 2010 Jan 20. PMID 20089307
- [Background] Pizzolorusso G, Turi P, Barlafante G, Cerritelli F, Renzetti C, Cozzolino V, D'Orazio M, Fusilli P, Carinci F, D'Incecco C. Effect of osteopathic manipulative treatment on gastrointestinal function and length of stay of preterm infants: an exploratory study. Chiropr Man Therap. 2011 Jun 28;19(1):15. doi: 10.1186/2045-709X-19-15. PMID 21711535
- [Background] Rubinstein SM, de Zoete A, van Middelkoop M, Assendelft WJJ, de Boer MR, van Tulder MW. Benefits and harms of spinal manipulative therapy for the treatment of chronic low back pain: systematic review and meta-analysis of randomised controlled trials. BMJ. 2019 Mar 13;364:l689. doi: 10.1136/bmj.l689. PMID 30867144
- [Background] Seffinger M.A. (2018). Foundation of osteopathic Medicine. Silva, R. M. V. da, & Sousa, A. V. C. de. (2020). Fase crônica da COVID-19: desafios do fisioterapeuta diante das disfunções musculoesqueléticas. Fisioterapia Em Movimento, 33, 2-4. https://doi.org/10.1590/1980-5918.033.ed02
- [Background] Steel A, Peng W, Sibbritt D, Adams J. Introducing national osteopathy practice-based research networks in Australia and New Zealand: an overview to inform future osteopathic research. Sci Rep. 2020 Jan 21;10(1):846. doi: 10.1038/s41598-020-57918-7. PMID 31964999
- [Background] Thomas P, Baldwin C, Bissett B, Boden I, Gosselink R, Granger CL, Hodgson C, Jones AY, Kho ME, Moses R, Ntoumenopoulos G, Parry SM, Patman S, van der Lee L. Physiotherapy management for COVID-19 in the acute hospital setting: clinical practice recommendations. J Physiother. 2020 Apr;66(2):73-82. doi: 10.1016/j.jphys.2020.03.011. Epub 2020 Mar 30. PMID 32312646
- [Background] Toledo, F. O., Junior, W. M., Speciali, J. G., & Sobreira, C. F. D. R. (2011). PND66 Cross-Cultural Adaptation and Validation of the Brazilian Version of the Fatigue Severity Scale (FSS). Value in Health, 14(7), A329-A330. https://doi.org/10.1016/j.jval.2011.08.532
- [Background] Tozzi P, Bongiorno D, Vitturini C. Low back pain and kidney mobility: local osteopathic fascial manipulation decreases pain perception and improves renal mobility. J Bodyw Mov Ther. 2012 Jul;16(3):381-391. doi: 10.1016/j.jbmt.2012.02.001. Epub 2012 Mar 3. PMID 22703751
- [Background] Wiersinga WJ, Rhodes A, Cheng AC, Peacock SJ, Prescott HC. Pathophysiology, Transmission, Diagnosis, and Treatment of Coronavirus Disease 2019 (COVID-19): A Review. JAMA. 2020 Aug 25;324(8):782-793. doi: 10.1001/jama.2020.12839. PMID 32648899
- [Background] World Health Organization (WHO). (2010). Benchmarks for training in traditional/complementary and alternative medicine: Benchmarks for Training in Osteopathy.
- [Background] Wu Y, Xu X, Chen Z, Duan J, Hashimoto K, Yang L, Liu C, Yang C. Nervous system involvement after infection with COVID-19 and other coronaviruses. Brain Behav Immun. 2020 Jul;87:18-22. doi: 10.1016/j.bbi.2020.03.031. Epub 2020 Mar 30. PMID 32240762